CLINICAL TRIAL: NCT00663624
Title: Management of Hyperglycemia in the Emergency Room: A Randomized Clinical Trial of a Subcutaneous Insulin Aspart Protocol Coupled With Rapid Initiation of Basal Bolus Insulin Prior to Hospital Admission Versus Usual Care
Brief Title: Management of Hyperglycemia in the ER: A Randomized Clinical Trial of a Subcutaneous Insulin Aspart Protocol Coupled With Rapid Initiation of Basal Bolus Insulin Prior to Hospital Admission Versus Usual Care
Acronym: NOVO ER
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding for the study at the Emory site
Sponsor: Emory University (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Dawn Smiley MD, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00008143; e8143
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Subcutaneous aspart insulin every 2 hours
  Interventions: Drug: aspart insulin
- Active Comparator (Placebo Comparator): Usual care as prescribed by the ED physicians
  Interventions: Drug: Usual care as prescribed by the ED physicians.

INTERVENTIONS:
Drug: aspart insulin — subcutaneous aspart insulin every 2 hours
  Arms: Experimental
Drug: Usual care as prescribed by the ED physicians. — Usual care can be oral anti-diabetic agents, subcutaneous insulin therapy or a combination of both. Subcutaneous insulin used for usual care could include NPH, 70/30 insulin, aspart insulin, regular insulin or insulin glargine
  Arms: Active Comparator

SUMMARY:
In the Emergency Department (ED), diabetes is commonly encountered as a secondary diagnosis and many patients with uncontrolled diabetes are admitted to the hospital after initial evaluation in the ED. Currently there are no guidelines in the US for the management of hyperglycemia in patients with diabetes during the duration of evaluation and treatment in the ED. It is known that high blood glucose levels in hospitalized patients with diabetes are associated with increased risk of medical complications. In this study, we hypothesize that a defined two-step approach to the management of high blood sugars with insulin injections initiated in the ED may decrease length of stay in the ED or hospital, improve clinical outcome and prevent some hospital complications. In the first phase, patients with diabetes admitted to the ED that have a high blood sugar (BG 200mg/dL) will be randomized to receive scheduled aspart or the usual care as dictated by the ED physicians. In the second phase, patients enrolled in the first phase that are subsequently admitted to the hospital will receive a combination of detemir and aspart insulin or usual care as dictated by the Admitting Medicine Team. Detemir is a long-acting insulin which is given subcutaneously (under the skin) once daily. Aspart is a rapid-acting insulin which is given subcutaneously several times a day and frequently before meals. Detemir and aspart insulins are approved for use in the treatment of patients with diabetes by the FDA. Usual care can be oral anti-diabetic agents, subcutaneous insulin therapy or a combination of both. Subcutaneous insulin used for usual care could include NPH, 70/30 insulin, aspart insulin, regular insulin or insulin glargine.

This investigator-initiated research will be conducted at Grady Memorial Hospital, Atlanta and at Rush University Medical Center, Chicago, IL. Dr. Smiley will serve as principal investigator at the Atlanta site. A total of 120 patients will be recruited at Grady and 120 patients at the Rush University Medical Center, Chicago, IL. This study is supported by Novo Nordisk.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all of the following criteria will be considered for enrollment into the study:
* Males or females between the ages of 18 and 80 years admitted to a general medical service.
* A known history of type 2 diabetes mellitus > 3 months, receiving diet management, any combination of oral antidiabetic agents (sulfonylureas, metformin, thiazolidinediones) and/or insulin therapy.
* Subjects must have an admission blood glucose > 140 mg and < 400 mg/dL and no evidence of ketoacidosis (serum bicarbonate < 18 mEq/L, venous or arterial pH < 7.30, positive serum or urinary ketones).

Exclusion Criteria:

* Subjects with increased blood glucose concentration, but without a known history of diabetes.
* Subsequent finding of diabetic ketoacidosis or hyperosmolar non-ketotic syndrome after initial evaluation.
* Patients with acute critical or surgical illness and/or expected to require admission to a critical care unit (ICU, CCU), or to undergo surgery during the hospitalization course.
* History of current drug or alcohol abuse.
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Inability to give informed consent
* Female patients who are pregnant or are breast feeding
* Patients who have clinically significant liver disease with ALT/AST > 3 X the upper range of normal
* Patients with serum creatinine ≥3.5 mg/dL for males or ≥ 3.0 mg/dL for females or currently treated with dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
to determine whether initiation of hyperglycemia management in the ED with scheduled aspart insulin for patients versus usual care with type 2 diabetes will result in a decrease in subsequent hospital length of stay. | once all subjects have been recruited

SECONDARY OUTCOMES:
to determine diff. in the mean BG during the ED stay, the mean BG achieved during hospital, frequency of hypoglycemia during the ED and hospital visits among those treated with the scheduled protocol insulin regimen vs. usual hyperglycemia mgmt | once all subjects have been recruited

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Smiley, MD, Principal Investigator — Emory SOM